CLINICAL TRIAL: NCT03464539
Title: Occult Obscure Gastrointestinal Bleeding (OGIB) in Colonic Diverticulitis Using Polyglucosamine: a Registry Study Following a Standard Management Protocol
Brief Title: Occult Obscure Gastrointestinal Bleeding
Acronym: OGIB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Blymum Srl (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20180206_UC
Record Dates: First submitted 2018-02-07; First posted 2018-03-14 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2018-02

CONDITIONS: Gastrointestinal Bleeding
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD patients (Other): PG low molecular weight chitosan 3 times per day
  Interventions: Dietary Supplement: PG low molecular weight chitosan

INTERVENTIONS:
Dietary Supplement: PG low molecular weight chitosan — The product 1000 mg of Polyglucosamine was administered three times per day before and in between main meals
  Other Names: Low molecular weight polyglucosamine

SUMMARY:
To test the activity of a polyglucosamine (PG) together with a Standard Management protocol (SM) on the occult and obscure gastrointestinal bleeding (OGIB) and the clinical symptoms in patients suffering from colonic diverticulitis (CD).

DETAILED DESCRIPTION:
The trial was conducted in a single center and subjects were participating to the San Valentino Vascular Screening Project (SVVSP). Sixty patients with history of colonic diverticulitis (CD) and occult obscure gastrointestinal bleeding (OGIB) were recruited. All subjects were following a Standard Management (SM) protocol consisting of diet and lifestyle modifications, and were freely choosing to be treated with polyglucosamine (PG) or to follow the SM only. Two groups of 30 cases each were formed and followed for 3 months.

Diet was controlled three times (baseline and during the first and third month), through the Food Intake Assessment (FIA) which consisted of the weekly analysis of 25 different servings (e,g fruits, vegetables, pulses, first dish, meat, processed meat, cheese). The lifestyle modification consisted of physical exercise (9 MET (Metabolic Equivalents) -h/week of brisk walking) and oral hygiene.

The main variable was OGIB, that was measured using Hemoccult Sensa Fecal Occult Blood Procedure.

Ancillary variables where the hs-CRP (high sensitivity C Ractive Protein) and the daily gastrointestinal discomfort (GID) measured thorough a visual analogue scale (VAS) from 0 to 10.

All variables were taken at baseline, after one and three months with the exception of GID that was measured also after one week of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged between 55 to 65 years (males and females).
* CD diagnosis.
* DICA (Diverticular Inflammation and Complication Assessment) class DICA 2 or DICA 3.
* OGIB positive to Hemoccult Sensa Fecal Occult Blood Procedure.

Exclusion Criteria:

* Subjects with Class DICA > 3.
* Therapy with mesalazine antibiotics and probiotics.
* Cancer of any type (a part from benign polyposis),
* Alcoholism.
* Parkinsonism.
* Alzheimer's Disease.
* Severe depression.
* Drug addiction.

Ages: 55 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-05-15 (Actual); Study Completion 2017-06-15 (Actual)

PRIMARY OUTCOMES:
Change of Occult bleeding | Baseline - 1 month - 3 months
  Bleeding in feces

SECONDARY OUTCOMES:
Gastrointestinal discomfort | Baseline - 1 week - 1 month - 3 months
  Measurement through visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Gianni Belcaro, MD, Study Director — University of Chieti
Locations (1):
- Spoltore - Pescara, Pescara, Italy

IPD SHARING:
Plan to Share IPD: No